CLINICAL TRIAL: NCT00925210
Title: Bronchoscopic Approach to the Peripheral Lung Nodule - An Alternative Approach Using Peripheral Endobronchial Ultrasonography and Electromagnetic Navigation Bronchoscopy
Brief Title: Bronchoscopic Approach to the Peripheral Lung Nodule - An Alternative Approach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: David R. Stather, University of Calgary
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22176
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Solitary Pulmonary Nodule; Lung Cancer
Keywords: Endobronchial ultrasound; Electromagnetic Navigation Bronchoscopy; Bronchoscopy; Ultrasonography
MeSH Terms: conditions — Solitary Pulmonary Nodule; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequential pEBUS - ENB (Experimental)
  Interventions: Procedure: Sequential pEBUS - ENB

INTERVENTIONS:
Procedure: Sequential pEBUS - ENB — Subject will undergo bronchoscopy with peripheral endobronchial ultrasonography to identify the peripheral lung nodule. If the lesion is identified with pEBUS, samples will be collected.
  If the lesion is not found by pEBUS, the electromagnetic navigation system will be deployed and directed to the lesion of interest, once again using pEBUS to confirm final location before samples are collected.

SUMMARY:
Patients presenting with solitary or multiple lung nodules often require tissue confirmation in order to guide further management and determine if the lesion is benign or malignant. Several bronchoscopic techniques have emerged which have significantly improved the diagnostic yield of bronchoscopy in this setting, and in particular the combination of peripheral Endobronchial Ultrasonography (pEBUS) and Electromagnetic Navigation Bronchoscopy (ENB) has resulted in diagnostic yields of nearly 90%. In an attempt to reduce the significant cost of this combined approach, the sequential use of pEBUS followed by the more costly ENB technique only if a lesion is not identified on the ultrasound image could be as accurate. This study aims to determine the diagnostic yield of this sequential approach in patients with lung nodule(s).

ELIGIBILITY:
Inclusion Criteria:

* Age >16 years
* Lung nodule (s) identified on CT scan
* Clinical decision to obtain tissue biopsy of lung lesion
* CT guided biopsy not preferred technique (previous negative CT guided biopsy or technically difficult nodule location or perceived high risk of pneumothorax or other complications)
* Pleural based lesion only if: Inaccessible by CT guided biopsy or previous CT guided biopsy non-diagnostic

Exclusion Criteria:

* Lack of informed consent
* Nodule less than 1 cm or greater than 6 cm long axis
* Mediastinal adenopathy >2cm short axis on CT chest
* Evidence of endobronchial abnormality on chest CT
* Medical contraindication to bronchoscopy
* Patients with lesions highly suspicious for lung cancer, potentially resectable with lobar or lesser resection and without significantly increased operative risk factors will not be entered into this study prior to surgical evaluation.
* Patient with implanted electronic medical device
* Uncontrolled or irreversible coagulopathy (platelets <100, INR >1.3, use of clopidogrel in the 7 days prior to bronchoscopy)
* Confirmed or suspected pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
diagnostic yield

SECONDARY OUTCOMES:
sensitivity, specificity, positive and negative predictive value
Impact of nodule size (<2 cm, 2-3 cm, >3cm) and distribution on diagnostic yield
Independent and incremental yield of BAL, biopsy, needle aspiration and brush cytology will be compared
Complication rate

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Foothills Medical Center, Calgary, Alberta
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec

REFERENCES:
- See also: Related Info — http://www.ucalgary.ca/ipm/